CLINICAL TRIAL: NCT00774163
Title: Phase 1: Safety of Lactobacillus Reuteri in Healthy Volunteers
Brief Title: Safety of Lactobacillus Reuteri in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Johns Hopkins Bloomberg School of Public Health (Other); Asociacion Benefica Prisma (Other)
Responsible Party: Principal Investigator, Richard A. Oberhelman, Professor, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDA IND# 13710; 1R01AT002733-01A1 (NIH)
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2013-07-12 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: probiotics; lactobacillus; reuteri; none (safety only)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period
  Interventions: Biological: Lactobacillus reuteri
- 2 (Placebo Comparator): Placebo oil preparation, administered as 5 drops of the oil vehicle used in manufacturing the Lr suspension, given once daily for a five-day study period
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Lactobacillus reuteri — Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period
  Other Names: BioGaia Probiotic Drops
  Arms: 1
Other: Placebo — 5 drops of the oil vehicle used in manufacturing the Lr suspension, given once daily for a five-day study period
  Arms: 2

SUMMARY:
This is a phase one study to assess the safety of daily dosing of Lactobacillus reuteri in healthy adults in Peru. It is conducted as a preliminary study in support of a clinical trial to assess safety and efficacy of Lactobacillus reuteri versus placebo for treatment of pediatric diarrhea in Peru.

DETAILED DESCRIPTION:
This is a phase I blinded randomized study of the safety and tolerability of Lactobacillus reuteri DSM 17938 given daily for a period of five consecutive days. Upon enrollment subjects will be randomized to one of two treatment groups in a ratio of treatment to placebo of 2:1. Subjects will be randomized to receive either:

A. Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period that corresponds to a dose of the closely related L. reuteri ATCC 55730 strain that has shown to be therapeutic for infantile colic. The strain used in this study (DSM 17938) has been cured of an antibiotic resistance plasmid found in the original BioGaia strain (L. reuteri ATCC 55730).

B. Placebo oil preparation, administered as 5 drops of the oil vehicle used in manufacturing the Lr suspension, given once daily for a five-day study period (BioGaia AB, Stockholm, Sweden).

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 with no exclusion criteria
* Subject is a male or, if the subject is female and of childbearing potential then she must have a negative serum or urine pregnancy test result within 48 hours of initiating study preparations and agree to use an acceptable method of contraception. Acceptable methods of contraception include depot forms of progesterone containing therapies or an intrauterine device (IUD).

Exclusion Criteria:

* No enrollment of family members in households where any of the following are present:

  * Another study participant in the household
  * Pregnancy or current breastfeeding by any household member
  * Presence of an infant under age 6 months living in the household
  * Presence of immune suppressed individuals or use of immunosuppressive agents (corticosteroids, methotrexate) by any household member
  * Presence of a serious congenital anomaly or chronic medical condition that would contraindicate participation in any household member, including history of gastrointestinal surgery, chronic gastrointestinal illness, abnormal intestinal anatomy, or abnormal bowel functionality
* Allergy to penicillin or cephalosporins
* History of antibiotic use in the last 30 days
* Use of probiotic products within the past 90 days
* History of diarrheal illness within the past 30 days
* Presence of fever or a pre-existing adverse event monitored in the study
* Positive results on serum diagnostic tests for antibodies to HIV, Hepatitis B core antigen, and Hepatitis C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Oberhelman, MD, Principal Investigator — Tulane School of Public Health and Tropical Medicine; Margaret N Kosek, MD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Community of Santa Clara, Iquitos, Loreto, Peru

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were inoformed of the study in community meetings in Santa Clara, Peru. Interested individuals were enrolled at the study clinic between Feb. 23, 2010 and April 2, 2010.
Groups:
- Lactobacillus Group: Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period
- Placebo Group: Placebo oil preparation, administered as 5 drops of the oil vehicle used in manufacturing the Lr suspension, given once daily for a five-day study period
Period: Overall Study
Arm/Group | Lactobacillus Group | Placebo Group
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Group | Placebo Group | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 15 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (2.0) | 32.3 (2.3) | 36.8 (1.8)
Gender [Count of Participants; unit: Participants]
  Female | 23 | 9 | 32
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Peru | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Blood Culture for L. Reuteri
Description: To assess association between administration of Lactobacillus reuteri (Lr) strain DSM 17938 and abnormal lab values (CBC, BUN, Creatinine, AST, ALT, blood culture).
Time Frame: participants were followed for an average of 36 days
Population: 2:1 randomization Lactbacillus:placebo using a randomizatin table as specified in the protocol
Measure: Number; unit: participants
Groups:
- Lactobacillus Reuteri Group: Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
participants | 0 | 0

2. Secondary Outcome: Number of Subjects With at Least One PCR Positive Stool Specimen
Time Frame: Average of 36 day follow up period
Measure: Number; unit: participants
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
participants | 9 | 5

3. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Vomiting Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: Days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (Days of observation) | 1230 | 615
days with symptom reported | 4 | 3

4. Primary Outcome: Mean Daily Temperature
Description: Measured daily during 5 days of study product administration
Time Frame: 5 days of study product administration
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Degrees Celcius | 36.02 (0.5) | 36.04 (0.5)

5. Primary Outcome: Leukocyte Count on Day 5
Time Frame: Measured on day 5
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
cells per cubic millimeter | 6936 (1331) | 7893 (1168)

6. Primary Outcome: Serum Alanine Aminotransferase (ALT) in Female Participants
Time Frame: Day 5
Population: limited to females
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 23 | 9
units per liter (U/L) | 30.3 (18.0) | 22.2 (12.4)

7. Primary Outcome: Serum ALT in Males
Time Frame: Day 5
Population: limited to males
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 7 | 6
units per liter (U/L) | 31.1 (29.7) | 27.8 (10.4)

8. Primary Outcome: Serum Aspartate Aminotransferase (AST) in Females
Time Frame: Day 5
Population: limited to females
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 23 | 9
units per liter (U/L) | 28.3 (13) | 22.4 (5.1)

9. Primary Outcome: Serum AST in Males
Time Frame: Day 5
Population: limited to males
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 7 | 6
units per liter (U/L) | 31 (16.1) | 31 (16.9)

10. Primary Outcome: Blood Urea Nitrogen
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
mg/dl | 22.4 (7.0) | 19.3 (5.4)

11. Primary Outcome: Serum Creatinine
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
mg/dl | 0.73 (0.16) | 0.73 (0.24)

12. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Pruritis Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (days of observation) | 1230 | 615
days with symptom reported | 1 | 12

13. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Headache Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (days of observation) | 1230 | 615
days with symptom reported | 67 | 32

14. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Malaise Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (days of observation) | 1230 | 615
days with symptom reported | 13 | 19

15. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Diarrhea Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (days of observation) | 1230 | 615
days with symptom reported | 18 | 5

16. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Myalgia Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (days of observation) | 1230 | 615
days with symptom reported | 41 | 15

17. Secondary Outcome: Clinical Tolerance of Lactobacillus Reuteri (Lr) Strain DSM 17938 Based on Number of Days With Subjective Fever Reported
Time Frame: Day 0 through 6 weeks after Day 0
Measure: Number; unit: days with symptom reported
Units Other Than Participants: days of observation
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Number analyzed (Participants) | 30 | 15
Number analyzed (days of observation) | 1230 | 615
days with symptom reported | 15 | 2

ADVERSE EVENTS:
Time Frame: 6 months from initiation of study
Description: AEs are scored as grade 1= mild, grade 1= moderate, grade 3 = severe, and grade 4 = life threatening based on the subject's interpretation of their symptom severity.
Arm/Group | Lactobacillus Reuteri Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 27/30 | 13/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus Reuteri Group (N=30) | Placebo Group (N=15)
Nausea and vomiting (Gastrointestinal disorders) | 5 (8) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 4 (4)
Headache (Nervous system disorders) | 20 (38) | 9 (23)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (13) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (7)
Fever (Infections and infestations) | 5 (6) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (13) | 6 (10)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 5 (7)
vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0)
dysuria (Renal and urinary disorders) | 6 (17) | 3 (7)
laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lumbar pain (Musculoskeletal and connective tissue disorders) | 15 (22) | 5 (9)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (4)
sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No